CLINICAL TRIAL: NCT03035903
Title: Energy Cost for Holding a MedGem® Indirect Calorimeter
Acronym: MEDGEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: WW International Inc (Industry)
Responsible Party: Principal Investigator, Eric Ravussin, Associate Executive Director for Clinical Science, Pennington Biomedical Research Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PBRC 2016-086
Record Dates: First submitted 2017-01-26; First posted 2017-01-30 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Resting Metabolic Rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Not holding, then holding the MedGem® (Experimental): Subjects will be seated in an armless chair and have a RMR measurement taken while not holding, then holding a MedGem® Indirect Calorimeter.
  Interventions: Device: Not holding, then holding the MedGem®; Device: Holding, then not holding the MedGem®
- Holding, then not holding the MedGem® (Active Comparator): Subjects will be seated in an armless chair and have a RMR measurement taken holding, then not holding a MedGem® Indirect Calorimeter.
  Interventions: Device: Not holding, then holding the MedGem®; Device: Holding, then not holding the MedGem®

INTERVENTIONS:
Device: Not holding, then holding the MedGem® — Subjects will have a RMR measurement taken first while not holding the MedGem®, and then while holding the MedGem®
Device: Holding, then not holding the MedGem® — Subjects will have a RMR measurement taken first while holding the MedGem®, and then while not holding the MedGem®

SUMMARY:
The goal of this clinical protocol is to perform a randomized crossover study to determine the energy cost of holding the MedGem® device above a person's normal resting metabolic rate (RMR) compared to not holding the MedGem® device.

DETAILED DESCRIPTION:
Forty (40) subjects will be randomized to two (2) RMR measurements separated by a 40-minute rest (washout) period. The two RMR evaluation periods are as follows:

1. RMR with MedGem® Indirect Calorimeter
2. RMR without MedGem® Indirect Calorimeter

Study recruitment will be performed at PBRC. Screening, consenting, and all study procedures will be performed within a single study visit at PBRC within the Inpatient Unit. All subjects will be introduced to the ventilated hood to determine presence of claustrophobia prior to enrollment (i.e., signing of the consent form).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65 y
* BMI 25-40 kg/m2

Exclusion Criteria:

* Diabetes mellitus
* Current smoker
* Presently on a weight loss regimen
* Medications: diabetes, oral steroids, blood pressure drugs, weight loss drugs
* Claustrophobia
* Pregnant or breastfeeding
* Congestive heart failure
* Chronic kidney disease
* Pacemaker or other metal implants

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Resting Metabolic Rate (RMR) | 3 hours
  Resting metabolic rate will be assessed via a DeltaTrac Metabolic Cart

CONTACTS AND LOCATIONS:
Overall Officials: Eric Ravussin, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No
The data will be not be shared outside of Weight Watchers and the Investigators listed on the protocol for this study.